CLINICAL TRIAL: NCT06710041
Title: Effects of Kinesiotaping in Carpal Tunnel Syndrome Treatment: a Randomized Controlled Trial
Brief Title: Kinesiotaping in Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Hanife BAYKAL ŞAHİN, Asistant Professor, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020/38
Record Dates: First submitted 2024-11-21; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Carpal Tunnel Syndrome (CTS)
Keywords: carpal tunnel syndrome; Kinesiotaping; Sham taping
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Athletic Tape; Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kinesiotaping plus tendon and nerve gliding exercises (Active Comparator): Kinesiotaping was applied 3 times with 5-day intervals
  Interventions: Device: Kinesiotape; Other: Exercise
- Sham taping plus tendon and nerve gliding exercises (Sham Comparator): Sham taping was applied 3 times with 5-day intervals without stretching and without having the proper position.
  Interventions: Other: Exercise; Device: sham taping
- tendon and nerve gliding exercises alone (Other): The control group received exercise therapy only
  Interventions: Other: Exercise

INTERVENTIONS:
Device: Kinesiotape — Kinesiotape, when applied with a specific method and tension, significantly reduces the pressure on the median nerve by extending the transverse carpal ligament. It regulates edema under the skin and improves lymphatic and blood circulation. It reduces muscle spasms, eases the movement of tendons and fascia, and reduces pain through neurological suppression
  Arms: Kinesiotaping plus tendon and nerve gliding exercises
Other: Exercise — Tendon and nerve gliding exercise
Device: sham taping — In the sham taping group, kinesiotape was applied with two I bands without stretching and without having the proper position. This group was considered as the placebo group.
  Arms: Sham taping plus tendon and nerve gliding exercises

SUMMARY:
Objective: Kinesiotaping (KT) is a relatively new technique, which reduces the pressure on the median nerve by extending the transverse carpal ligament. The aim of this study was to evaluate the effectiveness of KT on Carpal tunnel syndrome (CTS) in a randomized, placebo-controlled manner.

Methods: Patients were randomly divided into three groups: Group 1 (KT plus tendon and nerve gliding exercises), Group 2 (sham-taping plus exercises) and Group 3 (exercises alone, control group). KT was applied 3 times with 5-day intervals throughout the study, with "neural technique" for median and ulnar nerves and "area correction technique" for carpal tunnel releasing. In the placebo group kinesiotapes were applied without stretching and proper position. Hand grip strength, VAS, Boston Carpal Tunnel Syndrome Questionnaire (BCTQ), and Short Form-12 (SF-12) were measured as outcome parameters at the first visit, 3rd and 6th week.

ELIGIBILITY:
Inclusion Criteria:

* clicical diagnosis of mild and moderate CTS
* having the CTS symptoms for at least 6 weeks

Exclusion Criteria:

* electrophysiological diagnosis of severe CTS,
* thenar atrophy,
* local corticosteroid injection or KT application or physical therapy treatment for CTS within the last 3 months,
* patients with secondary metabolic causes for CTS (such as diabetes mellitus, pregnancy, rheumatoid arthritis, sarcoidosis, thyroid disease),
* patients with other conditions that may cause neck and arm pain (cervical disc hernia, arthritis, epicondylitis, rotator cuff syndrome),
* a history of fracture in the wrist,
* previous CTS surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
pain level | From enrollment to the end of treatment at 3 weeks
  pain level was assessed using visual analog scale.The minimum and maximum values were 0 and 10, and higher scores mean a better outcome.

SECONDARY OUTCOMES:
Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) | From enrollment to the end of treatment at 6 weeks
  The BCTQ is a disease specific questionnaire to evaluate the symptom severity and functional capacity. High scores indicate increased symtom severity and low functional capacity

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical University, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Geler Kulcu D, Bursali C, Aktas I, Bozkurt Alp S, Unlu Ozkan F, Akpinar P. Kinesiotaping as an alternative treatment method for carpal tunnel syndrome. Turk J Med Sci. 2016 Jun 23;46(4):1042-9. doi: 10.3906/sag-1503-4. PMID 27513402
- [Background] Giray E, Karali-Bingul D, Akyuz G. The Effectiveness of Kinesiotaping, Sham Taping or Exercises Only in Lateral Epicondylitis Treatment: A Randomized Controlled Study. PM R. 2019 Jul;11(7):681-693. doi: 10.1002/pmrj.12067. Epub 2019 Mar 28. PMID 30609278